CLINICAL TRIAL: NCT05672303
Title: The Effect of Grasp Reflex Stimulation on Pain During Vaccine Administration
Brief Title: Pain During Vaccine Administration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Collaborators: MSc Elif Simay KOÇ (Unknown)
Responsible Party: Principal Investigator, Türkan Kadiroğlu, Pricipal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: B.30.2.ATA.0.01.00/277
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Infant, Newborn, Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Routine procedure will be applied
- Experimental (Experimental): Palmar grasp reflex will be stimulated with routine procedure.
  Interventions: Behavioral: Palmar grasp reflex

INTERVENTIONS:
Behavioral: Palmar grasp reflex — The reflex can be stimulated by moving an object distally across the palm. In the study, at the beginning of the vaccine administration, the right hand of the infant will be moved distally along the palm with the researcher's index finger, thus providing reflex stimulation.
  Arms: Experimental

SUMMARY:
Many painful interventions that cause pain and stress are applied to preterm babies in the neonatal intensive care unit for diagnosis and treatment. In neonatal care and reduction of acute interventional pain; Non-pharmacological methods including behavioral, psychological and environmental regulations should be used.

In the hepatitis B vaccine administered to preterm babies, stimulating the grasping reflex can make the preterm baby feel safe and calm. In the literature, there are many studies aimed at reducing pain in preterm newborns. However, no study has been found on the effect of grasping reflex stimulation on pain and crying in hepatitis B vaccine administration to preterm infants.

This study was planned to examine the effect of grasping reflex on pain and crying duration in preterm infants with hepatitis B vaccine.

ELIGIBILITY:
Inclusion Criteria:

* 28-36 gestational week
* No congenital malformation
* follow up with a diagnosis of respiratory distress syndrome,
* receive oxygen support with a nasal cannula or tube,
* not receive mechanical ventilation support,
* no contraindications for hepatitis B vaccine administration,
* stable vital signs before vaccination,
* not receive analgesic sedation treatment
* whose parents give verbal and written consent to participate in the study.

Exclusion Criteria:

* Infants of parents who did not give informed voluntary consent will not be included in the study.
* Decreased oxygen saturation levels
* Tachycardia just before the vaccine administration
* Invasive intervention in the right hand.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-04-01 (Actual)

PRIMARY OUTCOMES:
pain level will be measured in the premature baby | 15 minutes
  PIPP-R Form: The PIPP scale, developed by Stevens et al. in 1996, is a validated assessment tool used to evaluate acute pain experienced by preterm infants during interventional procedures (Stevens et al., 1996). This scale was revised by Stevens et al. in 2014 (Stevens et al., 2014). The PIPP-R was adapted into Turkish in 2019 (Taplak, & Bayat, 2019). PIPP-R consists of behavioral subscales such as frowning, squeezing eyes, nasolabial furrow, physiological and behavioral status including heart rate and SPO2, and contextual subscales such as gestational age.

SECONDARY OUTCOMES:
Crying time | 15 minutes
  Crying time will be evaluated in seconds with a coronometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Türkan Kadiroğlu, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No